CLINICAL TRIAL: NCT02991079
Title: Effectiveness of a Multifactorial Intervention to Improve Diet and Physical Activity in Diabetic Patients From Primary Care: A Randomised Controlled Trial
Brief Title: Effectiveness of a Multifactorial Intervention to Improve Diet and Physical Activity in Diabetics From Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRS 1276/B/16
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Food Habits; Health education; Physical activity; Information and Communication Technologies
MeSH Terms: conditions — Feeding Behavior; Health Education; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Lifestyle counseling (Active Comparator): Counseling on physical activity and Mediterranean diet.
  Interventions: Other: Control: Lifestyle counseling
- Intervention group (Experimental): Add for three months a smartphone with an app (EVIDENT) to improve alimentation and physical activity, five cardio-health rides and feeding workshop.
  Interventions: Other: Intervention group; Other: Control: Lifestyle counseling

INTERVENTIONS:
Other: Intervention group — Smartphone with APP (EVIDENT) for 3 months, cardio-health rides and feeding workshop.
  Counseling on physical activity and Mediterranean diet.
  Arms: Intervention group
Other: Control: Lifestyle counseling — Conseling on physical activity and nutrition (intervention)

SUMMARY:
This is a randomized, clinical trial aimed at diabetics between 25-70 years (with no cardiovascular disease) selected at urban primary care health clinics in Salamanca (Spain). It is aimed at assessing the effects of adding an ICT (information and communication technology) tool, developed for the Smartphone application and group activities of healthy food and cardio-health rides in support of behavioral and educational recommendations in the increased physical activity and adaption to the Mediterranean dietary pattern.

DETAILED DESCRIPTION:
Objective:

The main objective of this study is to evaluate the effect of adding a multifactorial intervention (ICT tool for Smartphone, cardio-health rides and a standardized advice about eating habits) to the usual care in the increase of the physical activity, in order to reach the international recommendations and in the Increased adherence to the Mediterranean diet in type 2 diabetic patients. Secondary objectives will be to evaluate the effect of intervention in improving dietary patterns, cardiovascular risk factors and metabolic control.

Design and setting:

A randomised controlled clinical trial, with two parallel groups, aimed at assessing the effects of adding an ICT tool and group activities on healthy food and cardio-health rides (intervention), in support of behavioral and educational recommendations (control) in the increased physical activity and adaption to the Mediterranean dietary pattern.

Study setting:

Primary Care Health Area of Salamanca in the Research Unit of La Alamedilla, belonging to the Spanish Network for Preventive Activities and Health Promotion (redIAPP) and Salamanca Institute for Biomedical Research (IBSAL).

Study population:

200 patients with Diabetes Mellitus Type 2, aged between 25-70 years, of both sexes, who meet selection criteria and signed informed consent.

Each participant will make three visits: baseline, three and twelve months post-intervention.

Measuring the effect of the intervention:

The validated 14-point Mediterranean Diet Adherence Screener, the International Physical Activity Questionnaire (IPAQ), pedometer, laboratory values including glucose and glycosylated hemoglobin, and quality of life questionnaire (SF -12).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Diabetes Mellitus Type 2 since 25 to 70 years.

Exclusion Criteria:

* Older than 70 years are excluded, due to difficulties in the use of ICTs.
* History of cardiovascular events (acute myocardial infarction, stroke, etc).
* Diagnosis of clinically demonstrable neurological and/or neuropsychological disease.
* Muscular-skeletal pathology that inhibit mobility.
* Those with any other circumstance that the investigators consider could interfere with the study procedures.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-17 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet using the validated 14-point Mediterranean Diet Adherence Screener | 1 year
  Principal endpoint of alimentation, will be measured using the validated 14-point Mediterranean Diet Adherence Screener.
Self-reported physical activity measured by the International Physical Activity Questionary - Short Form | 1 year
  Measured by the International Physical Activity Questionary - Short Form

SECONDARY OUTCOMES:
Increase physical activity measurement by pedometer | 1 year
  Measurement by pedometer.
HbA1c | 1 year
  Measurement by laboratory test sampling
Fasting Plasma Glucose | 1 year
  Measurement by laboratory test sampling
Quality of life measured by SF-12 test | 1 year
  Measurement by SF-12 test
Cardiovascular risk factors measured by Framingham Risk Score | 1 year
  Measurement by Framingham Risk Score

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit - The Alamedilla Center for Health, Salamanca, Spain

REFERENCES:
- [Derived] Alonso-Dominguez R, Recio-Rodriguez JI, Patino-Alonso MC, Sanchez-Aguadero N, Garcia-Ortiz L, Gomez-Marcos MA. Acute effect of healthy walking on arterial stiffness in patients with type 2 diabetes and differences by age and sex: a pre-post intervention study. BMC Cardiovasc Disord. 2019 Mar 8;19(1):56. doi: 10.1186/s12872-019-1039-x. PMID 30849947
- [Derived] Alonso-Dominguez R, Patino-Alonso MC, Sanchez-Aguadero N, Garcia-Ortiz L, Recio-Rodriguez JI, Gomez-Marcos MA. Effect of a multifactorial intervention on the increase in physical activity in subjects with type 2 diabetes mellitus: a randomized clinical trial (EMID Study). Eur J Cardiovasc Nurs. 2019 Jun;18(5):399-409. doi: 10.1177/1474515119835048. Epub 2019 Feb 26. PMID 30808196
- [Derived] Alonso-Dominguez R, Gomez-Marcos MA, Patino-Alonso MC, Sanchez-Aguadero N, Agudo-Conde C, Castano-Sanchez C, Garcia-Ortiz L, Recio-Rodriguez JI. Effectiveness of a multifactorial intervention based on an application for smartphones, heart-healthy walks and a nutritional workshop in patients with type 2 diabetes mellitus in primary care (EMID): study protocol for a randomised controlled trial. BMJ Open. 2017 Sep 14;7(9):e016191. doi: 10.1136/bmjopen-2017-016191. PMID 28912193